CLINICAL TRIAL: NCT00577213
Title: Diagnosis of Hemangiomas and Vascular Malformations Using Non-invasive Imaging Devices
Brief Title: Diagnosis of Hemangiomas and Vascular Malformations
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 47573; Chancellor's Fund
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Hemangiomas; Vascular Malformations; Venular Malformations; Venous Malformations; Lymphatic Malformations; Arteriovenous Malformations
Keywords: Diagnosis; Hemangiomas; Vascular Malformations; Venular Malformations; Venous Malformations; Lymphatic Malformations; Arteriovenous Malformations
MeSH Terms: conditions — Hemangioma; Vascular Malformations; Lymphatic Abnormalities; Arteriovenous Malformations; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To develop a non-invasive, simple and affordable, measurement technique to differentiate hemangiomas from subtypes of VMS. The purpose of this study is to determine the best office based diagnositc instrument for differentiating the subtype of vascular lesions. The instrument must be simple and affordable so it can be used by primary car physicians in the doctor office. The procedure will be based on non-invasive and unharmful measurements that will be compared to the diagnosis from specialized physicians in this field and the final pathology.

ELIGIBILITY:
Inclusion Criteria:

* Suspected Hemangioma, Vascular Malformations (VMS) including venular Malformations (port-wine stain, PWS), Venous Malformations, Lymphatic Malformations, Arteriovenous Malformations or mixed malformations.

Exclusion Criteria:

* All pregnant individuals will be excluded, since physiologic changes of pregnancy could alter characteristics of the vascular lesion.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with vascular lesions from the patient populations at Arkansas Children's Hospital (ACH) and the University of Arkansas for Medical Sciences (UAMS) will be recruited for the study. Approximately 45 subjects from Arkansas Children's Hospital and approximately 10 subjects from the University of Arkansas for Medical Sciences will be recruited for a total of 55.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2007-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gal Shafirstein, Ph.D., Principal Investigator — UAMS, ACH, Central Arkansas Veterans Healthcare System; Jessica L Boswell, Study Director — UAMS, ACH, Central Arkansas Veterans Healthcare System